CLINICAL TRIAL: NCT02109120
Title: Dynamic Changes of MMP9 Concentration Cross Carotid Endarterectomy Monitoring Particulate Cerebral Embolisation
Brief Title: MMP-9 Monitoring Particulate Cerebral Embolisation
Acronym: MMP9MPCE
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-0321
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2013-09

CONDITIONS: Cerebral Embolic Damage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — serum,Freeze-saving -80℃
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- carotid endarterectomy (CEA): CEA patients with vein blood collection
  Interventions: Procedure: vein blood collection

INTERVENTIONS:
Procedure: vein blood collection — 5 ml peripheral vein blood samples were collected from each patient admitted to our study at the following time-points：Pre-operative（morning of surgery），just before declamping，30mins after declamping and post-operative（12h）.

SUMMARY:
1. In carotid endarterectomy(CEA) surgery, the dynamic changes of plasma MMP9 concentration cross CEA will be identified.
2. And the part of patients suffered particulate cerebral embolic injury, their MMP9 level will increase in the early stage after CEA.

ELIGIBILITY:
Inclusion Criteria:

-All patients enrolled had at least ≥70% unilateral or bilateral stenosis of Internal -Carotid Artery， or those who had a <70% stenosis but obvious cerebral ischema symptoms had been existed.

Exclusion Criteria:

* Exclusion criteria included poor temporal window
* Refused to cooperate with us
* Nonatheromatous such as takayasu arteritis and fibromuscular dysplasia.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients under CEA in the PUMCH
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
postoperative ischemic stroke | 7 days after surgery

SECONDARY OUTCOMES:
postoperative elevation of plasma MMP9 | perioperative phage

CONTACTS AND LOCATIONS:
Locations (1):
- vascular surgery department of PUMCH, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Molloy KJ, Thompson MM, Schwalbe EC, Bell PR, Naylor AR, Loftus IM. Elevation in plasma MMP-9 following carotid endarterectomy is associated with particulate cerebral embolisation. Eur J Vasc Endovasc Surg. 2004 Apr;27(4):409-13. doi: 10.1016/j.ejvs.2004.02.001. PMID 15015192
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed?term=Elevation+in+plasma+MMP-9+following+carotid+endarterectomy+is+associated+with+particulate+cerebral+embolisation&TransSchema=title&cmd=detailssearch